CLINICAL TRIAL: NCT00729976
Title: Oral Versus Rectal Ibuprofen for Fever in Young Children - a Randomized Control Study.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Eran Kozer, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 091/08
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2010-03

CONDITIONS: Fever
Keywords: Ibuprofen; Suppository; febrile children
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ibuprofen Suppository
  Interventions: Drug: Ibuprofen suppository
- 2 (Active Comparator): Ibuprofen suspension
  Interventions: Drug: Ibuprofen Suspension

INTERVENTIONS:
Drug: Ibuprofen suppository — 5-10mg/Kg of ibuprofen
  Arms: 1
Drug: Ibuprofen Suspension — 5-10mg/Kg
  Arms: 2

SUMMARY:
Fever is one of the most common symptoms in pediatrics and one of the most common reasons for visits in pediatricians' office and pediatric emergency departments. Many parents consider fever to be the most terrifying symptom.

Ibuprofen is an effective and safe treatment for febrile children. Until recently ibuprofen was available only in tablets suspension and as a liquid gel. All these dosage form are administered orally. Rectal suppositories are often essential for treating febrile children who cannot take medications by mouth (e.g vomiting). In the current study we aim to compare the effect on fever of ibuprofen given as suspension with ibuprofen suppositories.

ELIGIBILITY:
Inclusion Criteria:

Age: 3 mo- 4 years

* Weight 6 - 18 kg
* Rectal temperature > 38.50

Exclusion Criteria:

* Treatment with acetaminophen in the last 4 hours
* Treatment with Ibuprofen in the last 6 hours
* Unable to take oral or rectal medications
* Hypersensitivity to ibuprofen
* Renal failure
* Liver disease
* Rectal temperature can't be measured (due to anatomical or medical problem)
* Informed consent could not be granted

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Maximal change in temperature during the 4-hour period after enrollment. | 4 hours

SECONDARY OUTCOMES:
Proportion of patients with a drop of at least 1°C and 2°C in mean temperature at 4h. Decrement in fever at each time point, and the area under the temperature (versus time) curve. Proportion of patients with temperature < 38 at 4 hours. | 4 h

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel